CLINICAL TRIAL: NCT02057549
Title: Haloperidol vs Conventional Therapy for Gastroparesis
Acronym: HATGAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI left institution
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Carlos Roldan, MD, Associate professor in Emergency Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13040380
Record Dates: First submitted 2013-07-29; First posted 2014-02-07 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-07

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haloperidol plus Conventional Therapy (Experimental): Intravenous dose of haloperidol 5 mg in addition to conventional therapy. Conventional Therapy includes hydration via IV fluids, pain control with analgesics (usually opiates) frequently requiring multiple doses, also antiemetics (often requires multiple doses and different agents in attempts to control nausea and vomiting within this population), in addition to electrolytes abnormalities corrections as needed.
  Interventions: Drug: Haloperidol
- Conventional Therapy alone (Active Comparator): Conventional Therapy includes hydration via IV fluids, pain control with analgesics (usually opiates) frequently requiring multiple doses, also antiemetics (often requires multiple doses and different agents in attempts to control nausea and vomiting within this population), in addition to electrolytes abnormalities corrections as needed.
  Interventions: Drug: Conventional Therapy

INTERVENTIONS:
Drug: Haloperidol — Intravenous dose of haloperidol 5 mg.
  Other Names: Haldol
  Arms: Haloperidol plus Conventional Therapy
Drug: Conventional Therapy — Conventional Therapy includes hydration via IV fluids, pain control with analgesics (usually opiates) frequently requiring multiple doses, also antiemetics (often requires multiple doses and different agents in attempts to control nausea and vomiting within this population), in addition to electrolytes abnormalities corrections as needed.
  Arms: Conventional Therapy alone

SUMMARY:
Randomized controlled trial comparing haloperidol combined with conventional therapy and conventional therapy alone in patients with symptomatic gastroparesis.

DETAILED DESCRIPTION:
Study Design This study is a prospective, double-blind randomized placebo controlled trial involving adult emergency department (ED) patients who present with an acute exacerbation of gastroparesis. This study design will have two arms in the clinical trials. An experimental arm will receive an intravenous dose of haloperidol 5 mg in addition to conventional therapy, and the control arm will receive conventional therapy. Patients will be randomized as described below. Neither the physician nor the patient will be aware of the group to which the patient was randomized.

Methods Upon arrive at to the ED at the Memorial Hermann Hospital located in the Texas Medical Center; patients with gastroparesis (GP) exacerbation will be assessed for eligibility for enrollment in this trial by the clinicians on duty. Informed consent will be obtained from eligible patients that meet inclusion and exclusion criteria by trained ED residents. A 12 lead electrocardiogram will be performed to evaluate the presence of QT segment prolongation. Enrolled patients will be given 5 mg of intravenous haloperidol or equivalent volume of placebo pre-packaged and coded with a study ID number provided by the investigational pharmacy.

No unique identifiers or other PHI will be collected on enrolled patients. Information will also be recorded on the time elapsed from the time it took to provide the study medication and the time of the decision on disposition (admit or discharge). A record will be maintained if any additional medications including analgesics and antiemetics given to the patient before and after the study vial are given. Data will be collected on any adverse effects or complications the patients may experience (i.e. dystonic reactions, allergies etc.). After the data is collected at one hour for the primary outcome the trial will end and the physician will be unblended so they can choose subsequent medication.

All completed data collection forms will be dropped off in a secure locked mailbox and collected on a weekly basis by research staff. Collected forms will be housed in the ED office located in the Jesse Jones Library (JJL) 4th floor in a locked cabinet. Data will be entered electronically and analyzed using statistical package for the social sciences (SPSS) version 19.0. This database will be housed on a rights-protected research drive with limited access for viewing.

Informed Consent Patients will be notified of this study and they will be asked if they are interested in participating. If they are interested in participating, they will have the informed consent (IC) explained to them in either English or Spanish (Beaudoin, Nagdev, Merchant & Becker, 2010). The patient will sign, date, and put the time on the IC. The consenter will also do the same. A copy of the IC will be made in the ED and given to the patient for their records. The original copy will be housed in the regulatory binder located in JJL.

ELIGIBILITY:
Inclusion Criteria:

* Previous diagnosis of GP including those without formal gastric emptying studies.
* Patients presenting with unresolving nausea, vomiting, and abdominal pain that is attributable to their GP.

Exclusion Criteria:

* History of QT prolongation or presence on a 12 leads electrocardiogram.
* Presence of concomitant acute abdominal pathology including but not limited to hepatobiliary disease, ischemia, and abdominal aneurysm.
* Prisoners
* Hypotension (systolic blood pressure below 90 mm Hg)
* Pregnant women
* Patients who are cognitively impaired and/or unable to consent for the study
* Age <18
* Allergy to haloperidol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos J Roldan, MD, Principal Investigator — University of Texas
Locations (1):
- Lyndon Baines Johnson General Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roldan CJ, Chambers KA, Paniagua L, Patel S, Cardenas-Turanzas M, Chathampally Y. Randomized Controlled Double-blind Trial Comparing Haloperidol Combined With Conventional Therapy to Conventional Therapy Alone in Patients With Symptomatic Gastroparesis. Acad Emerg Med. 2017 Nov;24(11):1307-1314. doi: 10.1111/acem.13245. Epub 2017 Jul 26. PMID 28646590

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Started | 18 | 18
Completed | 15 | 18
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Continuous [Mean (Full Range); unit: years] | 47 [21 to 56] | 45 [20 to 57] | 46 [20 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 5 | 4 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief as Indicated by Number of Participants Not Requesting Additional Pain Medication
Time Frame: 1 hour after study medication given
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
Participants | 11 | 5

2. Secondary Outcome: Number of Participants Admitted to the Hospital After Emergency Department Visit
Time Frame: 2 hours after study medication given
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
Participants | 4 | 13

3. Secondary Outcome: Emergency Department Length of Stay (EDLOS)
Description: The "time frame" starts from the moment of receiving the study drug to the time when the decision for final disposition is made. Usually after symptoms are controlled, patients are given a PO challenge (food or drink) in order to establish if they are OK to go home. If symptoms return, additional medications are given, the treatment is consider failed and they are admitted to the Hospital.
  Patients will not be followed up if admitted to any service. The study ends when final disposition is made.
  Patients follow up after final disposition is not part of the study and will not be done.
Time Frame: at the time the decision for final disposition is made (about 8 hours)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
hours | 4.8 [4 to 10] | 9 [6.3 to 10.9]

4. Secondary Outcome: Pain Score as Measured by a Visual Analogue Scale (VAS)
Description: The Visual Analogue Scale (VAS) ranges from 0-10, with 0 being the absence of pain and 10 the worst imaginable pain.
Time Frame: before study medication given
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
units on a scale | 8.50 (1.82) | 8.28 (1.77)

5. Secondary Outcome: Pain Score as Measured by a Visual Analogue Scale (VAS)
Description: The Visual Analogue Scale (VAS) ranges from 0-10, with 0 being the absence of pain and 10 the worst imaginable pain.
Time Frame: 1 hour after study medication given
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
units on a scale | 3.13 (3.60) | 7.17 (2.81)

6. Secondary Outcome: Nausea Score as Measured by a Visual Analogue Scale (VAS)
Description: The Visual Analogue Scale (VAS) ranges from 1-5, with 1 being minimal nausea and 5 being severe nausea.
Time Frame: before study medication given
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
units on a scale | 4.53 (0.83) | 4.11 (0.96)

7. Secondary Outcome: Nausea Score as Measured by a Visual Analogue Scale (VAS)
Description: The Visual Analogue Scale (VAS) ranges from 1-5, with 1 being minimal nausea and 5 being severe nausea.
Time Frame: 1 hour after study medication given
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
units on a scale | 1.83 (1.92) | 3.39 (1.68)

8. Secondary Outcome: Nausea Relief as Indicated by Number of Participants Not Requesting Additional Antiemetic Medication
Time Frame: 1 hour after study medication given
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
Number analyzed (Participants) | 15 | 18
Participants | 11 | 13

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Haloperidol Plus Conventional Therapy | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 0/15 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No